CLINICAL TRIAL: NCT05769634
Title: Electrophysiologic Studies of Cognition in Epilepsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Allison Waters, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY-22-00529; R21MH126968-01A1 (NIH)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Drug-resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interoceptive Challenge Battery (Experimental): During simultaneous stereoelectroencephalography recording (n=20) patients will complete a series of three computer-based tasks designed to evoke changes in interoceptive attention and arousal.
  Interventions: Behavioral: Stereoelectroencephalography

INTERVENTIONS:
Behavioral: Stereoelectroencephalography — Computer-based tasks designed to evoke changes in interoceptive attention, arousal and anticipation will be completed. The first asks patients to attend to their heartbeat to manipulate interoceptive attention. The second asks patients to judge affective pictures to manipulate states of arousals. The third engages patients in a probabilistic reward-learning task, or gambling task, and anticipate the outcomes of risky decision-making. A final task guides patients to slow their breathing to 6 breaths per minute.

SUMMARY:
Interoception, or sensation from inside the body, is involved in a variety of clinical symptoms, such as tics, compulsions and negative mood. This study uses invasive recordings of brain activity and brain stimulation to better understand basic neural mechanisms of interoception and related behaviors. Outcomes of this study provide critical tools for future investigation into clinical symptoms that emerge from abnormal interoception.

DETAILED DESCRIPTION:
Abnormal interoceptive processing is observed across psychiatric and neurological conditions wherein core symptoms are motivated by diffuse bodily feeling: pervasive negative mood in Major Depression, compulsive urge in Obsessive Compulsive Disorder, urge to tic in Tourette Syndrome, and craving in addiction. Despite the prevalence of interoceptive abnormality, there is a scarcity of data on neurovisceral interactions in clinical populations. This knowledge gap can be attributed in part to a need for objective, neural measures of interoceptive processing. A candidate neural measure is the heartbeat evoked potential (HEP), a brain electrophysiological signal that is time-locked to the heartbeat and thought to index baroreceptor sensation in the chest cavity. While promising, basic characteristics of this signal are unknown, which limits its application to mechanistic and clinical research. Cortical sources of the HEP have been identified in the insula, yet spatial and temporal characteristics diverge across experimental paradigms. This suggests multiple functional correlates and cortical sources of the HEP index, including the insula. An added challenge is that the insula may be too deep for non-invasive recording and modulation, which necessitates invasive neural recording to explain non-invasive measures. Aim 1 validates neural source generators of the HEP with simultaneous invasive stereoelectroencephalography and dense array EEG on the scalp surface, while patients complete a battery of interoceptive tasks. Aim 2 investigates neural network dynamics during interoceptive attention, arousal and anticipation: theorizing that key clinical symptoms (e.g., tic, compulsions, negative mood) are learned behaviors in response to interoceptive cues, the research team tests the specific hypothesis that interoceptive activity is a predictor of reward-based decisions, particularly when decision-making demands a go with your gut strategy as reward outcomes are learned. Critically, Aim 3 then applies a deep breathing strategy to strategically perturb cardiac dynamics and disambiguate functional correlates of the HEP signal. Outcomes define properties of the HEP signal that must be known for this measurement strategy to inform and validate models of abnormal interoceptive circuit dynamics involving maladaptive responses to bodily distress.

ELIGIBILITY:
Inclusion Criteria:

* Epileptologists at Mount Sinai West have identified the patient as having drug-resistant epilepsy that may benefit from surgery
* Patient has or will undergo invasive monitoring as part of routine surgical management
* Patient has or will be implanted with a minimum of 6-8 bilateral SEEG pairs, including posterior and anterior insula, and at least four of the following targets:

  * ventral lateral prefrontal cortex
  * dorsal medial prefrontal cortex
  * mid-cingulate
  * subcallosal cingulate
  * amygdala
  * hippocampus
  * fusiform gyrus
* Sufficient use of hands to complete self-report questionnaires and tasks, as determined during pre-surgical neuropsychological assessment
* Normal or corrected to normal vision, determined by patient report
* Use of anti-epileptic drugs (AEDs) with known psychiatric complications will not be an exclusion criterion

Exclusion Criteria:

* Pre-operative neuropsychological testing indicates a Montreal Cognitive Assessment (MOCA) score < 26.
* English language proficiency insufficient to complete psychometric questionnaires and receive task instructions (<6th grade reading level) as determined by neuropsychologist at pre-operative assessment
* Vulnerable populations such as minors, pregnant women, cognitive impaired individuals and prisoners will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Waters, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to Allison.Waters@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included in the URL field below).
URL: https://labs.icahn.mssm.edu/waterslab/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interoceptive Challenge Battery
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Interoceptive Challenge Battery: During simultaneous stereoelectroencephalography recording (n=20) patients will complete a series of three computer-based tasks designed to evoke changes in interoceptive attention, arousal and anticipation.
  Stereoelectroencephalography: Three computer-based tasks designed to evoke changes in interoceptive attention, arousal and anticipation will be completed. The first asks patients to attend to their heartbeat to manipulate interoceptive attention. The second asks patients to judge affective pictures to manipulate states of arousals. A final task guides patients to slow their breathing to 6 breaths per minute.
Arm/Group | Interoceptive Challenge Battery
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 8
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Heartbeat Evoked Potential (HEP) for Attention
Description: The heartbeat evoked potential is a brain electrophysiological signal time locked to the "rpeak" of the cardiac signal and thought to reflect interoceptive sensation of baroreceptor firing in the chest cavity. The population average magnitude of the change in HEP following the experimental manipulation (mean, standard deviation, 95% confidence interval) will be reported.
Time Frame: 15 minutes
Measure: Mean (95% Confidence Interval); unit: µV
Arm/Group | Interoceptive Challenge Battery
Number analyzed (Participants) | 20
µV | -1.5 [-2.9 to -0.1]

2. Primary Outcome: Heartbeat Evoked Potential (HEP) for Arousal
Description: as for outcome 1
Time Frame: 15 minutes
Measure: Mean (95% Confidence Interval); unit: µV
Groups:
- Interoceptive Challenge Battery: During simultaneous stereoelectroencephalography recording (n=20) patients will complete a series of three computer-based tasks designed to evoke changes in interoceptive attention and arousal.
  Stereoelectroencephalography: Computer-based tasks designed to evoke changes in interoceptive attention, arousal and anticipation will be completed. The first asks patients to attend to their heartbeat to manipulate interoceptive attention. The second asks patients to judge affective pictures to manipulate states of arousals. A final task guides patients to slow their breathing to 6 breaths per minute.
Arm/Group | Interoceptive Challenge Battery
Number analyzed (Participants) | 20
µV | -2.02 [-3.15 to -0.89]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 15-minute period of stereoelectroencephalography recording.
Arm/Group | Interoceptive Challenge Battery
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT05769634/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT05769634/ICF_001.pdf